Protocol: version 3, 18/11/2015

The Acute effect of food structure on post prandial glucose

and subsequent metabolic responses

Statistical analysis

Statistical calculations were performed using SPSS software (version

21.0, SPSS Inc., Chicago, IL, USA), Microsoft Office Excel 2007 and

GraphPad Prism software (Prism 6.03, GraphPad Software Inc., CA,

USA).

The Shapiro-Wilk test was used to check the normality of the data  $(p \ge 1)$ 

0.01). Data were expressed as mean  $\pm$  the standard error of the mean

(SEM), unless otherwise stated. In cases of non-parametric data, log

transformation was performed before carrying out parametric statistical

tests. Time series data were analysed using repeated measures analysis

of variance (ANOVA) with post hoc Fisher LSD tests. Rheological data

compared using paired t-tests; P = 0.05 was considered statistically

significant.